CLINICAL TRIAL: NCT03351257
Title: Linked Color Imaging vs White-light Colonoscopy in the Characterization of Small and Diminutive Colon Polyps
Brief Title: The Characterization of Small and Diminutive Colonic Polyps in LCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 307LCI-DCPs
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Small Colon Polyps; Linked Color Imagimg; Diminutive Colon Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation of surface patterns and colors of polyps — examination of the surface patterns and colors of polyps using Linked color imaging and white-light

SUMMARY:
Colorectal cancer is a maior cause of morbidity and mortality worldwide.Colonoscopy and removal of all adenomas is the most efficient method to prevent colorectal cancer.The most colorectal polyps detected are small(<10mm) and diminutive(≦5mm) during colonoscopy.At that size,the are overwhelmingly hyperplastic or adenomatous,and rarely harbour high-grade dysplasia,cancer or sessile serrated adenoma/polyp.Traditional white-light endoscopy cannot reliably distinguish between small adenomatous and hyperplastic polyps,thus,real-time recognition of the polyp histology during colonoscopy has the potential to minimize both the costs and complications associated with endoscopic biopsy and polpectomy.Linked color imaging(LCI),a new system for endoscopy modality,creates clear and bright endoscopic images by using short-wavelength narrow-band laser light combined with white laser light on the basis of magnifying blue laser imaging(BLI) technology. it is easier to recognize a slight difference in color of the mucosa. This is a study to investigate the impact of Linked color imaging endoscopes on the in vivo histology prediction of colonic polyps.

DETAILED DESCRIPTION:
This is a prospective study comparing the accuracy of linked color imaging(LCI) and standard white light colonoscopes in the diagnosis of small and diminutive colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

- 1.ability to provide written informed consent and undergoing colonoscopy. 2.The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic work-up.

3.detection and retrieval for histologic examination of at least one polyp< 10mm in size and/or 5mm in size

Exclusion Criteria:

* Patients were previous colon resection
* Patients were a diagnosis of inflammatory bowel disease,familial polyp syndromes or poor bowel preparation
* suspected chronic stricture potentially precluding complete colonoscopy
* Patients had polypectomy or had coagulopathy/thrombocytopenia
* Patients had diverticulitis or toxic megacolon;previous radiation therapy to the abdomen or pelvis;severe cardiovascular,pulmonary,liver,or renal disease;and coagulation disorders or use of anticoagulants.
* all of polyps could influence surface pattern or/and color assessment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients who were referred for elective outpatient colonoscopy will be asked to enroll into this trial if the candidate meets the study inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
the accuracy of predicted in vivo polyp histology | 5 months
  the accuracy of predicted in vivo polyp histology

SECONDARY OUTCOMES:
Sensitivity | 5 months
  Sensitivity of white light endoscopy in predicting histology
specificity | 5 months
  sensitivity of white light endoscopy in predicting histology
Sensitivity | 5 months
  Sensitivity of LCI endoscopy in predicting histology

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Longcroft-Wheaton G, Brown J, Cowlishaw D, Higgins B, Bhandari P. High-definition vs. standard-definition colonoscopy in the characterization of small colonic polyps: results from a randomized trial. Endoscopy. 2012 Oct;44(10):905-10. doi: 10.1055/s-0032-1310004. Epub 2012 Aug 14. PMID 22893132
- [Background] Repici A, Hassan C, Radaelli F, Occhipinti P, De Angelis C, Romeo F, Paggi S, Saettone S, Cisaro F, Spaander M, Sharma P, Kuipers EJ. Accuracy of narrow-band imaging in predicting colonoscopy surveillance intervals and histology of distal diminutive polyps: results from a multicenter, prospective trial. Gastrointest Endosc. 2013 Jul;78(1):106-14. doi: 10.1016/j.gie.2013.01.035. Epub 2013 Apr 11. PMID 23582472
- [Background] Lee CK, Lee SH, Hwangbo Y. Narrow-band imaging versus I-Scan for the real-time histological prediction of diminutive colonic polyps: a prospective comparative study by using the simple unified endoscopic classification. Gastrointest Endosc. 2011 Sep;74(3):603-9. doi: 10.1016/j.gie.2011.04.049. Epub 2011 Jul 18. PMID 21762907
- See also: diminutive colonic polyps — https://www.ncbi.nlm.nih.gov/pubmed/26448409